CLINICAL TRIAL: NCT01029470
Title: A Multicentre, Prospective, Open Study to Describe the Effects of rhLH Supplement in Women With Hyporesponse to rFSH After Pituitary Downregulation.
Brief Title: To Describe the Effect of rhLH Supplementation in Women With Hyporesponse to rhFSH After Pituitary Downregulation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Chongqing Medical Center for Women and Children (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Jie Qiao, Peking University Third Hospital Reproductive Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR700642-606
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2009-12-10 (Estimated); Status verified 2009-12

CONDITIONS: Infertility
Keywords: Luveris; hyporesponse; pituitary downregulation; IVF; Infertility women
MeSH Terms: conditions — Infertility | interventions — Luteinizing Hormone, beta Subunit; follitropin alfa; Ovidrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Luveris (Experimental): Those subjects who experience hyponresponse to FSH stimulation during mid-follicle phase after pituitary downregulation will receive Luveris 75IU or 150IU IH injection daily till HCG day.
  Interventions: Drug: Luveris

INTERVENTIONS:
Drug: Luveris — Luveris 75IU or 150IU depending on the patient conditions, subcutaneous injection, Qd, from Day 8 till hCG Day
  Other Names: Gonal-f, ovidrel

SUMMARY:
Primary objective:

To evaluate the efficacy in terms of oocyte retrieval number of rLH supplement in women with hyporesponse to rFSH after pituitary downregulation.

Secondary objective:

To further explore the efficacy of rLH supplement in women with hyporesponse to rFSH after pituitary downregulation To evaluate the safety of rLH supplementation in hyporesponse women

DETAILED DESCRIPTION:
Primary endpoint:

Number of oocyte retrieved

Secondary endpoints:

1. Oestrodial on hCG day (pg/ml)
2. Number of embryos
3. Implantation rate (%)
4. Clinical pregnancy rate (%)
5. Ongoing PR per IVF cycle (%)
6. Abortion rate (%)
7. Ampoules of rFSH
8. FertiQoL score Safety endpoint: adverse events

ELIGIBILITY:
Inclusion Criteria:

1. 20-40 years old women
2. With menstrual cycles ranged 24-35 days, intraindividual variability±3 days
3. Basal FSH <10 IU/L at cycle D2-D5
4. 18 < BMI < 30
5. Presence of two ovaries
6. No ovarian stimulation over the past 3 months
7. Signed inform consent form.

Exclusion Criteria:

1. Polycystic ovarian syndrome
2. rAFS stage Ⅲ-Ⅳ endometriosis
3. Chromosomal abnormalities, endocrinological and/or autoimmune disorders.
4. More than two previously unsuccessful IVF.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-10 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Number of oocyte retrieved | 2009Dec-2010Oct

SECONDARY OUTCOMES:
1. Oestrodial on hCG day (pg/ml) Safety: adverse events | 2009 Dec-2010 Oct
2. Number of embryos | 2009 Dec-2010 Oct
3. Implantation rate (%) | 2009 Dec-2010 Oct
4. Clinical pregnancy rate (%) | 2009 Dec-2010 Oct
5. Ongoing PR per IVF cycle (%) | 2009 Dec-2010 Oct
6. Abortion rate (%) | 2009 Dec-2010 Oct
7. Ampoules of rFSH | 2009 Dec-2010 Oct
8. FertiQoL score Safety: adverse events | 2009 Dec-2010 Oct

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, MD, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University third Hospital, Beijing, Beijing Municipality, China